CLINICAL TRIAL: NCT05279404
Title: Effect of Electroacupuncture at Neiguan on Cardiac and Gastric Function
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: China Medical University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CMUH110-REC2-211
Record Dates: First submitted 2022-01-24; First posted 2022-03-15 (Actual); Last update posted 2022-03-15 (Actual); Status verified 2022-03

CONDITIONS: Cardiac and Gastric Function
MeSH Terms: interventions — Electroacupuncture; Acupuncture Therapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A - electroacupuncture (Experimental): electroacupuncture group Insert stainless steel acupuncture needles into Neiguan (cathode) and Jianshi (anode) on both sides and twist the needles.
  After that, the electroacupuncture machine was connected and 2 Hz electrical stimulation was administered for 30 minutes.
  The stimulation intensity was mainly based on slight muscle contractions and no pain in the subjects. At this time, cardiac function and electrogastrogram were recorded at the same time.
  Interventions: Other: electroacupuncture
- Group B - Sham electroacupuncture (Sham Comparator): Sham electroacupuncture group The method was the same as that of the electroacupuncture group, but the needles were only acupuncture under the skin of Neiguan and Jianshi without twisting the needles. The electroacupuncture machine was connected but no electrical stimulation was administered.
  Interventions: Other: electroacupuncture

INTERVENTIONS:
Other: electroacupuncture — Electroacupuncture at Neiguan and Jianshi acupoint
  Other Names: acupuncture

SUMMARY:
Acupuncture have been used in clinical treatment of diseases for at least 3,000 years, and the efficacy of acupuncture has been recognized by countries all over the world. However, most of the selected points for acupuncture treatment of diseases are based on ancient books or inheritance of experience. For example, the " Shizong Acupoint Ballad " of acupuncture records: "Neiguan (PC6) care about the chest and stomach", that is, acupuncture Neiguan can be used to treat chest, heart and stomach diseases. However, there is no scientific evidence to verify this argument so far that the Shizong Acupoint Ballad mentions "Neiguan care for the chest and stomach", and that means that Neiguan acupoint can treat the diseases of cardiovascular system and gastrointestinal system. The purpose is to verify the argument of "Neiguan care about the chest and stomach", and design a clinical trial of the Neiguan and Jianshi (PC5) on both sides of the electroacupuncture (EA) to simultaneously evaluate the heart and stomach functions. We designed a crossover test; total 72 subjects randomly equally divide the into a sham group (sham electroacupuncture) and an EA group [2Hz EA (PC6 is cathode) and PC5 is anode]. At least one week of washing time, then the EA group changed to a sham group and the sham group changed to an EA group.

In this study, it is expected that the EA at PC6 and PC5 will affect the heart function and the function of the stomach at the same time, verifying the argument that "the PC6 care of the chest and stomach" recorded in the Shizong Acupoint Ballad.

ELIGIBILITY:
Inclusion Criteria:

* (1) Normal and healthy participants
* (2) Male or female
* (3) The age range is 20 to 40 years old.
* (4) Those who participates and signs informed consent after explaining the research purpose and process in detail.

Exclusion Criteria:

* (1) Those with serious diseases, such as heart failure, chronic failure or cancer patients, etc.
* (2) Those who are allergic to stainless steel needles for acupuncture.
* (3) Pregnant or breastfeeding
* (4) Those who are taking medicines or food such as coffee, etc. that will affect heart function such as heart rate, or gastric peristalsis.
* (5) Unable to cooperate with researchers such as mental instability.
* (6) Those who do not sign the consent form.

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Estimated)
Dates: Start 2022-04-15 (Estimated); Primary Completion 2022-12-01 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Cardiac Function | thirty minutes.
  Evaluation of cardiac function with the "Osypka" non-invasive cardiac output monitor before electroacupuncture interventions .
  Cardiac function (OSCAR, non-invasive cardiac output meter) is first recorded for 30 minutes, and then intervention (electroacupuncture) is implemented, and cardiac function is recorded at the same time.
Cardiac Function | thirty minutes.
  Evaluation of cardiac function with the "Osypka" non-invasive cardiac output monitor during electroacupuncture interventions.
  Cardiac function (OSCAR, non-invasive cardiac output meter) is first recorded for 30 minutes, and then intervention (electroacupuncture) is implemented, and cardiac function is recorded at the same time.
Cardiac Function | thirty minutes.
  Evaluation of cardiac function with the "Osypka" non-invasive cardiac output monitor after electroacupuncture interventions.
  Cardiac function (OSCAR, non-invasive cardiac output meter) is first recorded for 30 minutes, and then intervention (electroacupuncture) is implemented, and cardiac function is recorded at the same time.
Cardiac Function | thirty minutes.
  After at least one week (washing time), the two groups would be switched, and cardiac function is measured once in the same pattern.
  Evaluation of cardiac function with the "Osypka" non-invasive cardiac output monitor before sham electroacupuncture interventions.
  Cardiac function (OSCAR, non-invasive cardiac output meter) is first recorded for 30 minutes, and then intervention (sham electroacupuncture) is implemented, and cardiac function is recorded at the same time.
Cardiac Function | thirty minutes.
  After at least one week (washing time), the two groups would be switched, and cardiac function is measured once in the same pattern.
  Evaluation of cardiac function with the "Osypka" non-invasive cardiac output monitor during sham electroacupuncture interventions.
  Cardiac function (OSCAR, non-invasive cardiac output meter) is first recorded for 30 minutes, and then intervention (sham electroacupuncture) is implemented, and cardiac function is recorded at the same time.
Cardiac Function | thirty minutes.
  After at least one week (washing time), the two groups would be switched, and cardiac function is measured once in the same pattern.
  Evaluation of cardiac function with the "Osypka" non-invasive cardiac output monitor after sham electroacupuncture interventions.
  Cardiac function (OSCAR, non-invasive cardiac output meter) is first recorded for 30 minutes, and then intervention (sham electroacupuncture) is implemented, and cardiac function is recorded at the same time.
Gastric Function | thirty minutes.
  Evaluation of gastric electrical rhythm with electrogastrography before electroacupuncture interventions.
  Gastric function (electrogastrography) is first recorded for 30 minutes, and then intervention (electroacupuncture) is implemented, and gastric function is recorded at the same time.
Gastric Function | thirty minutes.
  Evaluation of gastric electrical rhythm with electrogastrography during electroacupuncture interventions.
  Gastric function (electrogastrography) is first recorded for 30 minutes, and then intervention (electroacupuncture) is implemented, and gastric function is recorded at the same time.
Gastric Function | thirty minutes.
  Evaluation of gastric electrical rhythm with electrogastrography after electroacupuncture interventions.
  Gastric function (electrogastrography) is first recorded for 30 minutes, and then intervention (electroacupuncture) is implemented, and gastric function is recorded at the same time.
Gastric Function | thirty minutes.
  After at least one week (washing time), the two groups would be switched, and cardiac function is measured once in the same pattern.
  Evaluation of gastric electrical rhythm with electrogastrography before electroacupuncture and sham electroacupuncture interventions.
  Gastric function (sham electroacupuncture) is first recorded for 30 minutes, and then intervention (sham electroacupuncture) is implemented, and gastric function is recorded at the same time.
Gastric Function | thirty minutes.
  After at least one week (washing time), the two groups would be switched, and cardiac function is measured once in the same pattern.
  Evaluation of gastric electrical rhythm with electrogastrography during electroacupuncture and sham electroacupuncture interventions.
  Gastric function (sham electroacupuncture) is first recorded for 30 minutes, and then intervention (sham electroacupuncture) is implemented, and gastric function is recorded at the same time.
Gastric Function | thirty minutes.
  After at least one week (washing time), the two groups would be switched, and cardiac function is measured once in the same pattern.
  Evaluation of gastric electrical rhythm with electrogastrography after electroacupuncture and sham electroacupuncture interventions.
  Gastric function (sham electroacupuncture) is first recorded for 30 minutes, and then intervention (sham electroacupuncture) is implemented, and gastric function is recorded at the same time.

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) would be protected.